CLINICAL TRIAL: NCT05919108
Title: Neoadjuvant Neratinib in Stage I-III HER2-Mutated Lobular Breast Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Puma Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Laura Kennedy, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC-NCBRE23172; NCI-2023-04468 (Registry Identifier: NCI, Clinical Trials Reporting Program); 1R01CA273246-01A1 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer; Anatomic Stage II Breast Cancer; Anatomic Stage III Breast Cancer; Invasive Breast Lobular Carcinoma
MeSH Terms: conditions — Carcinoma, Lobular | interventions — neratinib; Magnetic Resonance Spectroscopy; Mastectomy, Segmental; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (endocrine therapy) (Active Comparator): Patients receive standard of care endocrine therapy over 4 weeks for 1 cycle. Patients undergo breast tissue biopsy during the lead-in window/cycle 1. Patients then endocrine therapy and neratinib PO daily for 20 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo breast surgery during weeks 24-25. Patients undergo collection of blood samples every 4 weeks while on treatment, at weeks 4 and 24, and at time of surgery. Patients undergo mammogram, ultrasound, or breast MRI prior to surgery.
  Interventions: Procedure: Endocrine Therapy; Procedure: Biopsy of breast; Drug: Neratinib; Procedure: Biospecimen Collection; Procedure: Mammogram; Procedure: Magnetic Resonance Imaging; Procedure: Breast Surgery
- Treatment B (endocrine therapy, neratinib) (Experimental): Patients receive standard of care endocrine therapy and neratinib PO over 4 weeks for 1 cycle. Patients undergo breast tissue biopsy during the lead-in window/cycle 1. Patients then continue endocrine therapy and neratinib PO daily for 20 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo breast surgery during weeks 24-25. Patients undergo collection of blood samples every 4 weeks while on treatment, at weeks 4 and 24, and at time of surgery. Patients undergo mammogram, ultrasound, or breast MRI prior to surgery.
  Interventions: Procedure: Endocrine Therapy; Procedure: Biopsy of breast; Drug: Neratinib; Procedure: Biospecimen Collection; Procedure: Mammogram; Procedure: Magnetic Resonance Imaging; Procedure: Breast Surgery; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Endocrine Therapy — Undergo endocrine therapy
Procedure: Biopsy of breast — Undergo breast biopsy
Drug: Neratinib — Taken by mouth
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Mammogram — Undergo Mammogram
Procedure: Magnetic Resonance Imaging — Undergo breast Magnetic Resonance Imaging
Procedure: Breast Surgery — Undergo Breast Surgery
Procedure: Ultrasound — Undergo Ultrasound
  Arms: Treatment B (endocrine therapy, neratinib)

SUMMARY:
This phase II trial tests how well neratinib prior to the primary treatment (neoadjuvant) works in treating patients with stage I-III HER2 mutated lobular breast cancers. Neratinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving neratinib in addition to normal therapy may work better in treating cancer than the endocrine therapy patients would normally receive.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine efficacy of neoadjuvant neratinib in combination with endocrine therapy.

SECONDARY OBJECTIVES:

I. Determine additional efficacy outcomes of neoadjuvant neratinib in combination with endocrine therapy.

II. Compare the safety and tolerability of neratinib plus endocrine therapy.

CORRELATIVE OBJECTIVE:

I. Establish HER2-mutant invasive lobular carcinoma (ILC) organoids.

OUTLINE: Patients are randomized to 1 of 2 treatments.

TREATMENT A: Patients receive standard of care endocrine therapy over 4 weeks for 1 cycle. Patients undergo breast tissue biopsy during the lead-in window/cycle 1. Patients then endocrine therapy and neratinib orally (PO) daily for 20 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo breast surgery during weeks 24-25. Patients undergo collection of blood samples every 4 weeks while on treatment, at weeks 4 and 24, and at time of surgery. Patients undergo mammogram, ultrasound, or breast magnetic resonance imaging (MRI) prior to surgery.

TREATMENT B: Patients receive standard of care endocrine therapy and neratinib PO over 4 weeks for 1 cycle. Patients undergo breast tissue biopsy during the lead-in window/cycle 1. Patients then continue endocrine therapy and neratinib PO daily for 20 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo breast surgery during weeks 24-25. Patients undergo collection of blood samples every 4 weeks while on treatment, at weeks 4 and 24, and at time of surgery. Patients undergo mammogram, ultrasound, or breast MRI prior to surgery.

After completion of study treatment, patients are followed up for 4 weeks after study drugs interruption.

ELIGIBILITY:
Inclusion Criteria:

Each patient will be entered into this study only if all of these criteria are met:

* Subjects aged 18 years or older at signing of informed consent.
* New diagnosis of clinical stage I-III HR+ histologically-proven (i.e. absent or decreased e-cadherin expression) invasive lobular carcinoma
* Synchronous breast tumors are permitted as long as the synchronous tumor is ER+ and HER2-negative.
* ER+ disease defined as ≥1% estrogen receptor (ER) positive consistent with current American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) or European Society of Medical Oncology (ESMO) guidelines)
* At the time of screening, histologically confirmed cancers in patients with previously documented activating HER2 mutation (see Appendix A) confirmed by a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalent laboratory.
* Archival tissue availability (if not available a fresh tumor biopsy will be required) and subject must agree to submission of sample for central testing
* Minimum tumor size of ≥1.5 cm by US, mammogram, MRI imaging, or clinical breast exam
* ECOG performance status 0 or 1
* Patients must have adequate hematologic, hepatic, and renal function. All laboratory tests must be obtained within 1 month of study entry. This includes:

  * Estimated glomerular filtration rate of ≥50 mL/min
  * Albumin ≥ 2.5 g/dL
  * ANC ≥1500/mm^3
  * Platelet count ≥100,000/mm^3
  * HgB ≥ 9 g/dL
  * Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
  * AST and ALT ≤ 3 x ULN
* Pre-, peri-, or post-menopausal, confirmed by history or laboratory testing as needed
* Diagnostic biopsy tissue availability with sufficient tumor to permit NGS (if not available, a fresh biopsy will be required)
* No prior treatment for current diagnosis of breast cancer
* For patients who are not postmenopausal (women) or surgically sterile (absence of ovaries and/or uterus or vasectomy), agreement to remain abstinent or to use two adequate methods of contraception (e.g., condoms, diaphragm, vasectomy/vasectomized partner, tubal ligation), during the treatment period and for at least 30 days after the last dose of study treatment. Hormone based oral contraceptives are not allowed on study. Postmenopausal is defined as:

  * Age ≥ 55 years
  * Age ≤ 55 years and amenorrheic for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression; or follicle stimulating hormone and estradiol in the postmenopausal range. Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception that has a low user dependency consistently and correctly.

Note: The effects of neratinib on the developing fetus are unknown and endocrine therapy is contraindicated in pregnancy. For this reason and because teratogenic effects have been observed in nonclinical studies and neratinib, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study participation, and for 1 month after the last dose of study medication. Should a woman become pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation and 3.5 months after completion of study treatment.

Exclusion Criteria:

* Evidence of distant metastatic disease
* Synchronous breast cancer that is estrogen receptor negative OR HER2-amplified OR requires treatment with neoadjuvant chemotherapy per the judgement of the treating physician
* Patients harboring ineligible somatic HER2 mutations, such as those that are subclonal in nature or those resulting in the expression of truncated proteins including alterations that result in premature stop codon or a change in reading frame (ie, frame shift mutations).
* Prior endocrine therapy for breast cancer within the last 2 years
* Women who are pregnant, are planning to become pregnant, or are breast-feeding
* Any investigational treatment for the current diagnosis of breast cancer
* HER2 amplification by FISH (HER2:CEP17 ratio >2.0) or IHC (HER2 (3+)
* Hepatic function impairment as defined by AST or ALT > 3x ULN OR total serum bilirubin > 1.5 (in patients with known Gilbert syndrome, a total bilirubin of > 3.0 x ULN or direct bilirubin > 1.5 x ULN)
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (eg, Crohn's disease, malabsorption, or Grade ≥2 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 4.0 [CTCAE version 4.0] diarrhea of any etiology at baseline.
* Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that could, in the Investigator's judgment, make the patient inappropriate for this study.
* Known hypersensitivity to any component of the investigational product, required combination therapy, or loperamide.
* Unable or unwilling to swallow tablets.
* Unable or unwilling to complete study procedures such as research biopsies or imaging
* Any medical condition that in the judgement of the co-investigator would impair the patient's ability to complete the planned study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative endocrine prognostic index score | Up to 5 years

SECONDARY OUTCOMES:
Pathological complete response rate | Up to 5 years
  Will be summarized for the entire cohort by response.
Change in Ki67 | At 4 weeks
Residual cancer burden index | Up to 5 years
  Will be summarized for the entire cohort by response
Rates of breast conservation therapy | Up to 5 years
  Will be summarized for the entire cohort by response
Incidence of adverse events (NCI Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kennedy, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (5):
- United States (5):
  - Emory University/ Winship Cancer Institute, Atlanta, Georgia
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas, Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT05919108/ICF_000.pdf